CLINICAL TRIAL: NCT07021495
Title: A Prospective, Multi-Center, Observational Biomarker Real-World Evidence Study for In-Depth Profiling of Patients With Chronic Immune-Mediated Inflammatory Skin Diseases in Daily Practice
Brief Title: SKIN Disease Profiling by an Exploratory, pRospective, Biomarker Study in dermatoloGY Practice (SKINERGY)
Acronym: SKINERGY
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Radboud University Medical Center (Other); Amsterdam University Medical Center (Other); UMC Utrecht (Other); Maastricht University Medical Center (Other); University Medical Center Groningen (Other); Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Principal Investigator, Prof. dr. Robert Rissmann, Prof. dr. Robert Rissmann, Leiden University Medical Center
Other Study IDs: SKINERGY; NWA.1389.20.182 (Other Grant/Funding Number: Dutch Research Council (NWO)); NGID (Other Grant/Funding Number: Next Generation ImmunoDermatology consortium)
Record Dates: First submitted 2025-05-20; First posted 2025-06-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Spontaneous Urticaria (CSU); Hidradenitis Suppurativa (HS); Psoriasis (PsO); Atopic Dermatitis (AD); CTCL/ Mycosis Fungoides
Keywords: Urticaria; Hives; Mast cells; Autoimmune; Autoallergic; Wheals; Angioedema; Abscess; Nodules; Sweat glands; Acne inversa; Eczema; Itchy, dry skin; Mycosis Fungoides; Skin patches; Tumors; T-cells; Lupus; Skin rash; Photosensitivity; Plaques; Scaling; Erythema; Induration; Inflammatory skin diseases; Immune-mediated; Deep phenotyping; Multi-omics; Transcriptomics; Lipidomics; Metabolomics; Proteomics; Genomics; Microbiomics; Imaging mass cytometry (CyTOF); Real-world practice; Standard care; NextGenerationImmunoDermatology; NGID; Biomarkers
MeSH Terms: conditions — Chronic Urticaria; Hidradenitis Suppurativa; Psoriasis; Dermatitis, Atopic; Mycosis Fungoides; Urticaria; Angioedema; Abscess; Eczema; Pruritus; Neoplasms; Exanthema; Photosensitivity Disorders; Plaque, Amyloid; Erythema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples (including blood sample for genomics analysis, optionally)
  * Skin punch biopsies (optional)
  * Tape strips of skin surface
  * Swab of skin surface
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (18):
- AD - CsA: Adult patients with moderate-to-severe AD who start treatment with cyclosporine A. Cyclosporine A (CsA) is a lipophilic, cyclic undecapeptide produced by fungi, acting as a potent immunosuppressant by inhibiting T-cell receptor activation. It's prescribed twice daily at 3-5 mg/kg/day, starting with 3 mg/kg/day and increasing based on clinical response. CsA inhibits cytokine production, especially interleukin-2 (IL-2). In the Netherlands, CsA is the only oral immunosuppressant for moderate-to-severe atopic dermatitis (AD). CsA has shown superiority over placebo in numerous trials, and is the treatment of choice for severe AD. Common adverse reactions include renal dysfunction, tremor, hirsutism, hypertension, diarrhea, nausea, and vomiting. Contraindications include hypersensitivity and certain drug combinations. Regular monitoring is necessary due to potential risks like acute infections, hepatotoxicity, and renal toxicity.
- AD - Anti-IL4/13: Adult patients with AD who start treatment with anti-IL4/13 (dupilumab, tralokinumab, lebrikizumab). Dupilumab is a human monoclonal antibody that targets the IL-4 receptor alpha chain, inhibiting IL-4 and IL-13. In the Netherlands, it's the first biologic registered for moderate-to-severe atopic dermatitis (AD). Administered subcutaneously every other week at 300mg, following a loading dose of 600mg at baseline, it follows standard treatment guidelines with regular monitoring. Dupilumab's efficacy has been shown in clinical trials, with long-term benefits in AD. Common adverse reactions include injection site reactions, conjunctivitis, arthralgia, oral herpes, and eosinophilia. Tralokinumab, another monoclonal antibody, neutralizes IL-13 to reduce AD symptoms. Administered similarly to dupilumab, its efficacy has also been demonstrated in trials, showing superiority over placebo. Common ADRs include upper respiratory infections, injection site reactions, and conjunctivitis.
- AD - JAK1 inhibitor: Adult patients with AD who start treatment with JAK1 inhibitors (upadacitinib/abrocitinib). Upadacitinib and abrocitinib are selective JAK1 inhibitors that reduce immune system activity by blocking Janus Kinases, enzymes involved in inflammatory responses, which drive atopic dermatitis (AD) symptoms like eczematous skin lesions and pruritus. Upadacitinib is dosed at 15mg or 30mg once daily, with clinical trials showing significant improvements in IGA-AD, EASI 75, and pruritus compared to placebo. Common ADRs include upper respiratory infections, acne, and herpes simplex. Abrocitinib is dosed at 100mg or 200mg once daily, with 200mg recommended for severe AD. It has also shown significant efficacy in clinical trials. ADRs for abrocitinib include nausea, headache, and acne.
- PSO - Anti-TNF: Adult patients with moderate-to-severe PSO who start treatment with anti-TNF (e.g. adalimumab, certolizumab, biosimilars). Adalimumab is a monoclonal antibody used to treat moderate-to-severe rheumatoid arthritis, plaque psoriasis, and hidradenitis suppurativa. It inhibits TNF, reducing inflammation. Common adverse events include infections, injection site reactions, headache, and musculoskeletal pain. For plaque psoriasis, the recommended dose is 80 mg at week 0, followed by 40 mg biweekly. Certolizumab, another TNF inhibitor, treats plaque psoriasis with an initial dose of 400 mg at weeks 0, 2, and 4, followed by 200 mg biweekly (or 400 mg if efficacy is insufficient).
- PSO - anti-IL23: Adult patients with moderate-to-severe PSO who start treatment with anti-IL 23 (e.g. guselkumab, risankizumab, tildrakizumab). Guselkumab (Tremfya) is an anti-IL-23 monoclonal antibody approved for moderate-to-severe plaque psoriasis in patients eligible for systemic treatment. It blocks IL-23 interaction with its receptor, reducing pro-inflammatory cytokines. The recommended dose is 100 mg at weeks 0 and 4, followed by 100 mg every 8 weeks. Common adverse reactions include respiratory tract infections and diarrhea. Risankizumab (Skyrizi) also targets IL-23, with a dosing regimen of 150 mg at weeks 0 and 4, followed by 150 mg every 12 weeks. Common AEs include respiratory infections, injection site reactions, tinea, headache, itching, fatigue, and rash. Tildrakizumab (Ilumetri) targets the IL-23 p19 subunit. It is dosed at 100 mg at weeks 0 and 4, followed by 100 mg every 12 weeks. Common AEs include respiratory infections, injection site pain, nausea, diarrhea, and headache.
- PSO - anti-IL17: Adult patients with moderate-to-severe PSO who start treatment with anti IL-17 (e.g. secukinumab, ixekizumab, brodalumab, bimekizumab). Secukinumab is an IL-17A inhibitor for psoriasis and hidradenitis suppurativa. It blocks IL-17 interaction with its receptor. The dose is 300 mg at weeks 0, 1, 2, 3, and 4, followed by 300 mg monthly. Common AEs include respiratory infections, nasopharyngitis, oral herpes, diarrhea, headache, and fatigue. Ixekizumab, another IL-17A inhibitor, is dosed at 160 mg in week 0, followed by 80 mg every 2 weeks for 10 weeks, then 80 mg every 4 weeks. AEs include injection site reactions and respiratory infections. Brodalumab binds IL-17RA, with a dose of 210 mg at weeks 0, 1, and 2, followed by biweekly doses. Common AEs include infections, tinea, headache, and fatigue. Bimekizumab inhibits IL-17A, IL-17F, and IL-17A/F, dosed at 320 mg at weeks 0, 4, 8, 12, and 16, followed by 320 mg every 8 weeks. Common AEs include infections, candidiasis, and fatigue.
- PSO - anti-TYK2: Adult patients with moderate-to-severe PSO who start treatment with TYK2 inhibitor (e.g. deucravacitinib). Deucravacitinib is a selective TYK2 inhibitor used for moderate-to-severe plaque psoriasis. It selectively binds the allosteric pocket of TYK2, leading to high selectivity in inhibition. Inhibiting TYK2 interferes with cytokine signaling involved in plaque psoriasis. The recommended dose is 6 mg daily. The most common adverse reactions occurring in ≥1% of patients are (viral) upper respiratory infections, nasopharyngitis, pharyngitis, sinusitis, herpes simplex, oral ulceration, acneiform rash, folliculitis, and increased creatine kinase levels.
- HS - anti-TNF: Adult patients with moderate-to-severe HS who start treatment with anti-TNF (e.g. adalimumab, certolizumab, biosimilars). Adalimumab is a monoclonal antibody used to treat moderate-to-severe rheumatoid arthritis, plaque psoriasis, and hidradenitis suppurativa. It inhibits TNF, reducing inflammation. Common adverse events include infections, injection site reactions, headache, and musculoskeletal pain. For hidradenitis suppurativa, the dose starts with 160 mg at week 0, then 80 mg at week 2, followed by 40 mg weekly or 80 mg biweekly.
- HS - anti-IL17: Adult patients with moderate-to-severe HS who start treatment with anti-IL 17, i.e. secukinumab, bimekizumab* (*once approved and reimbursed in the Netherlands). Secukinumab is an IL-17A inhibitor for psoriasis and hidradenitis suppurativa. It blocks IL-17 interaction with its receptor. The dose is 300 mg at weeks 0, 1, 2, 3, and 4, followed by 300 mg monthly. Common AEs include respiratory infections, nasopharyngitis, oral herpes, diarrhea, headache, and fatigue. Ixekizumab, another IL-17A inhibitor, is dosed at 160 mg in week 0, followed by 80 mg every 2 weeks for 10 weeks, then 80 mg every 4 weeks. AEs include injection site reactions and respiratory infections. Brodalumab binds IL-17RA, with a dose of 210 mg at weeks 0, 1, and 2, followed by biweekly doses. Common AEs include infections, tinea, headache, and fatigue. Bimekizumab inhibits IL-17A, IL-17F, and IL-17A/F, dosed at 320 mg at weeks 0, 4, 8, 12, and 16, followed by 320 mg every 8 weeks. Common AEs include infections, cand
- MF - Topical chlormethine: Adult patients with stage 1 or 2 cutaneous T-cell lymphoma subtype mycosis fungoides who start treatment with topical chlormethine. Chlormethine (CL) gel 0.016% (Ledaga®) is an FDA-approved orphan drug (since August 23, 2013) for stage IA and IB mycosis fungoides in patients previously treated with skin-directed therapy. It forms DNA interstrand crosslinks, blocking replication and transcription, leading to cell death in rapidly dividing cells.
  CL gel showed no systemic absorption up to 6 hours post-application and after 1 month (Lessin et al., 2013). In a follow-up study with CL gel 0.04%, no detectable drug or degradation product was found in blood up to 6 months (Kim et al., 2014).
  In a randomized trial (n=128, median 52 weeks), 61.7% had skin-related side effects, mainly dermatitis (54.7%), pruritus (20.3%), infections (11.7%), ulceration/blistering (6.3%), and hyperpigmentation (5.5%). Hypersensitivity occurred in 2.3%. No systemic side effects or overdoses were reported.
- MF - Topical corticosteroids: Adult patients with stage 1 or 2 cutaneous T-cell lymphoma subtype mycosis fungoides who start treatment with topical corticosteroids. Topical corticosteroids are anti-inflammatory medications that are used in the treatment of various inflammatory skin diseases, such as cutaneous T-cell lymphoma subtype mycosis fungoides. Corticosteroids inhibit the release of inflammation factors and therefore, the inflammatory response is reduced. Topical corticosteroids are divided in four subclasses, based on their potency. Topical corticosteroids are generally described as highly effective in the treatment of certain skin diseases. The recommended dose of topical corticosteroids depends on the subclass and specific therapy, however, generally 2 applications per day are recommended over a limited time period. AE's as skin thinning, and increased risk of infections are often reported.
- MF - PUVA/UB-B: Adult patients with stage 1 or 2 cutaneous T-cell lymphoma subtype mycosis fungoides who start treatment with PUVA/UV-B. Psoralen UV-A (PUVA) is used to treat cutaneous T-cell lymphoma subtype mycosis fungoides. It combines UVA light with psoralen, a drug that makes the skin more sensitive to light. Typically, 2-3 treatments per week are required for effectiveness. Common side effects include nausea (due to psoralen) and skin redness (from UVA). Long-term use may lead to premature skin aging.
  UV-B light therapy, including narrowband UVB, is also used for (folliculotropic) mycosis fungoides. It uses short-wave UVB light that penetrates the outer skin layers. While generally safer than older phototherapies, long-term treatment may increase the risk of skin cancer.
- CSU - anti-IgE: Adult patients with moderate to severe CSU who start (add-on) treatment with anti-IgE. Omalizumab is a highly effective treatment for chronic spontaneous urticaria. It is a recombinant humanized IgG1 monoclonal antibody targeting immunoglobulin E (IgE). Experimental models in cynomolgus monkeys and mice have been used to study its pharmacokinetics. The mouse model focused on antigen-independent behavior in the absence of IgE binding. After subcutaneous administration, bioavailability was 90% in mice and 64-104% in monkeys. Peak concentrations occurred around day 5, with a half-life of approximately 7 days. Clearance of omalizumab:IgE complexes was significantly slower than that of free IgE, leading to up to 20-fold increases in total IgE levels.
  In use since 2004, omalizumab has a well-established safety profile in asthma, CSU, and CRSwNP, both in trials and post-marketing. The most common AEs in CSU include nasopharyngitis, headache, sinusitis, and injection site reactions.
- CSU - CsA: Adult patients with moderate to severe CSU who start (add-on) treatment with cyclosporin A. Cyclosporine A (CsA) is a lipophilic, cyclic undecapeptide produced by fungi, acting as a potent immunosuppressant by inhibiting T-cell receptor activation. It's prescribed twice daily at 3-5 mg/kg/day, starting with 3 mg/kg/day and increasing based on clinical response. CsA inhibits cytokine production, especially interleukin-2 (IL-2). In the Netherlands, CsA is the only oral immunosuppressant for moderate-to-severe atopic dermatitis (AD). CsA has shown superiority over placebo in numerous trials, and is the treatment of choice for severe AD. Common adverse reactions include renal dysfunction, tremor, hirsutism, hypertension, diarrhea, nausea, and vomiting. Contraindications include hypersensitivity and certain drug combinations. Regular monitoring is necessary due to potential risks like acute infections, hepatotoxicity, and renal toxicity.
- CSU - anti-BTK: Adult patients with moderate to severe CSU who start (add-on) treatment with anti-BTK*. Bruton's tyrosine kinase (BTK) inhibitors block BTK, a key enzyme in B-cell receptor signaling that controls B-cell activation and survival. By inhibiting BTK, these drugs disrupt B-cell function and pathological immune responses.
  They are mainly approved for B-cell cancers like chronic lymphocytic leukemia (CLL) and mantle cell lymphoma (MCL). Common BTK inhibitors include ibrutinib, acalabrutinib, and zanubrutinib, which are orally administered and generally well tolerated.
  BTK also plays a crucial role in mast cell and basophil activation via the FcεRI receptor, central to chronic spontaneous urticaria (CSU). Inhibiting BTK blocks mast cell degranulation and histamine release, reducing symptoms in CSU patients, especially those unresponsive to antihistamines or omalizumab. This makes BTK inhibitors promising oral therapies for CSU.
  *once approved and reimbursed in the Netherlands
- CLE - Topical corticosteroids: Adult patients with mild to severe chronic lupus erythematosus (CLE) who start treatment with topical corticosteroids. Topical corticosteroids are anti-inflammatory medications that are used in the treatment of various inflammatory skin diseases, such as cutaneous T-cell lymphoma subtype mycosis fungoides. Corticosteroids inhibit the release of inflammation factors and therefore, the inflammatory response is reduced. Topical corticosteroids are divided in four subclasses, based on their potency. Topical corticosteroids are generally described as highly effective in the treatment of certain skin diseases. The recommended dose of topical corticosteroids depends on the subclass and specific therapy, however, generally 2 applications per day are recommended over a limited time period. AE's as skin thinning, and increased risk of infections are often reported.
- CLE - Hydroxychloroquine: Adult patients with mild to severe chronic lupus erythematosus (CLE) who start treatment with HCQ. HCQ is an antimalarial used to treat rheumatoid arthritis, systemic lupus erythematosus, and cutaneous lupus. It accumulates in lysosomes, raising pH, and inhibits TLR3, TLR7, and TLR9, reducing plasmacytoid dendritic cell activation and lowering IFNα and TNF production. HCQ also suppresses T and B cell activation, reducing Th1, Th2, and Th17 responses, while sparing cytotoxic T cells.
  Orally, HCQ has 74% bioavailability, a Tmax of 2-4.5 hours, and a plasma half-life around 32 days. It concentrates in blood cells and tissues like lungs, kidneys, and eyes. Metabolized in the liver, it is cleared by the kidneys.
  Common side effects are nausea, abdominal pain, and diarrhea, often reduced by taking HCQ with food. Risks include hypoglycemia, retinopathy, cardiac toxicity, and blood count changes, requiring regular monitoring.
- CLE - Methotrexate: Adult patients with mild to severe chronic lupus erythematosus (CLE) who start treatment with methotrexate. Methotrexate (MTX), introduced in 1947 for cancer, has been used since the 1980s at low doses to treat rheumatoid arthritis (RA). It is given once weekly, orally or by injection (s.c., i.m., i.v.).
  MTX's anti-inflammatory effects involve inhibition of nucleotide synthesis, NF-κB signaling, JAK-STAT pathway modulation, nitric oxide production, adenosine release, and regulation of certain RNAs.
  Orally, MTX has ~70% bioavailability with peak levels in 1-2 hours; subcutaneous administration offers higher and faster plasma levels. About 50% binds serum proteins and accumulates in liver, kidneys, and spleen as polyglutamates. The half-life varies from 3 to 17 hours.
  Common side effects include nausea, fatigue, mouth sores, liver enzyme elevation, and leukopenia. Early detection allows reversibility; patients are closely monitored. Folic acid is recommended to reduce adverse events.

SUMMARY:
The goal of this observational study is to comprehensively profile six immune-mediated inflammatory diseases, including atopic dermatitis (AD), plaque psoriasis (PSO), hidradenitis suppurativa (HS), cutaneous T-cell lymphoma subtype mycosis fungoides (MF), chronic spontaneous urticaria (CSU), and cutaneous lupus erythematosus (CLE) in daily practice. Data will be compared with data from healthy volunteers. This study is part of the larger NGID (Next Generation ImmunoDermatology) initiative, of which the main objective is to develop infrastructure that enables personalised patient care. The main questions the SKINERGY study aims to answer are:

* Which biomarkers can discriminate between responders and non-responders to treatment in patients with AD, CLE, CSU, HS, MF, and PSO?
* How do disease-related biomarkers in patients with AD, CLE, CSU, HS, MF, and PSO differ from those in healthy volunteers?
* Which (multi-omics) biomarkers are associated with disease subtypes and predict response or non-response to (targeted) therapies in daily clinical practice?
* How do biomarker profiles compare across different cohorts of patients with immune-mediated inflammatory skin diseases (AD, CLE, CSU, HS, MF, PSO)
* How do biomarker levels change over time in response to treatment in these patient populations?
* Which skin tissue biomarkers are associated with disease progression or treatment response?
* How do the genomic profiles of patients differ across diseases or correlate with treatment outcomes?
* Can additional imaging biomarkers enhance the characterization of disease profiles or treatment monitoring over time?

Researchers will compare both differences beween patients within a disease group in different treatment arms, as well as patients within the same treatment arm. Additionally, biomarker profiles of patients with different diseases will be evaluated. These comparisons will be made to see if shared or distinct biomarker patterns exist across diseases and treatments, which could inform patient stratification, optimize therapeutic decision-making, and identify potential targets for future interventions.

Participants will start medication according to national guidelines for the treatment of their inflammatory skin disease (AD: Cyclosporin A, anti-IL4/13, or anti-JAK; PSO: anti-TNF, anti-IL23, ani-IL17, anti-TYK2; HS: anti-TNF, anti-IL17; MF: CHLORM, TSC, PUVA-UV-B; CSU: anti-IgE, Cyclosporin A, anti-BTK*; CLE: TSC, HCQ, MTX)

*once approved and reimbursed in the Netherlands

Participants will:

* Take the prescribed medication for their skin disease (in line with standard care in the Netherlands).
* Visit the clinic for a study visit combined with their standard care appointment 3 times (baseline, month 3, and month 6. An additional 4th visit at month 12 is optional).
* Fill in an online set of questionnaires from home, 3 times during the study period (an additional 4th time is optional).
* Patients with CSU fill in the UAS7 (and if applicable the AAS7) daily for the study period.

DETAILED DESCRIPTION:
Atopic dermatitis (AD), cutaneous lupus erythematosus (CLE), chronic spontaneous urticaria (CSU), hidradenitis suppurativa (HS), cutaneous T-cell lymphoma (CTCL, subtype mycosis fungoides, MF), and plaque psoriasis (PSO) are diverse immune-mediated inflammatory skin diseases with complex and often poorly understood pathophysiologies. Genetic, immunological, and environmental factors contribute variably across these conditions, leading to heterogeneous clinical presentations. Despite advances, the identification and validation of specific biomarkers remain limited, hampering precise diagnosis, disease subtyping, and treatment response prediction. For example, AD involves epidermal barrier defects and immune dysregulation; CLE features autoimmune mechanisms and diverse clinical subtypes; CSU results from mast cell activation; HS is driven by follicular occlusion and chronic inflammation; CTCL involves malignant T-cell proliferation in the skin; and PSO is characterized by immune-driven keratinocyte hyperproliferation. The Next Generation ImmunoDermatology project aims to address these challenges by deeply profiling these diseases to discover biomarkers that define disease endotypes and predict therapy response, ultimately enabling personalized treatment strategies.

The investigations will profile various aspects of the disease, including patient-reported outcomes, the clinician-reported outcomes, biophysical, imaging, cellular, microbiological, molecular, blood-based and tissue biomarkers.

This multicenter, open-label, longitudinal biomarker study follows 720 patients with six inflammatory skin diseases-AD, PSO, HS, CSU, CLE, and MF-for one year after starting standard-of-care treatment. Multimodal data are collected at baseline, 3, 6, and 12 months. An additional 120 healthy controls are included for baseline comparison and followed for 6 weeks. Each disease includes multiple treatment arms (N=40 per arm):

* AD: cyclosporine A; anti-IL-4/13 (dupilumab, tralokinumab, lebrikizumab); JAK1 inhibitors (upadacitinib, abrocitinib)
* PSO: anti-IL-23 (guselkumab, risankizumab, tildrakizumab); anti-IL-17 (secukinumab, ixekizumab, brodalumab, bimekizumab); anti-TNFα (adalimumab, certolizumab); TYK2 inhibitor (deucravacitinib)
* HS: anti-TNFα (adalimumab); anti-IL-17 (secukinumab, bimekizumab*)
* MF: topical chlormethine; topical corticosteroids; phototherapy (PUVA/UV-B)
* CSU: anti-IgE (omalizumab*); cyclosporine A; BTK inhibitors* (remibrutinib, rilzabrutinib)
* CLE: topical corticosteroids; hydroxychloroquine; methotrexate

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Able to understand and provide a written informed consent prior to any study procedures
2. Male or non-pregnant female, ≥18 years of age
3. Patient is willing to refrain from extensively washing (including bathing, swimming) the target lesional skin 12 hours before every study visit day.
4. Patient is willing and able to comply with the study protocol
5. Female participants are willing to not get pregnant between M0 until M12, from study entry to the last study visit
6. The patient is willing to start the prescribed treatment.

Disease-specific inclusion criteria

For patients with AD:

To be eligible to participate in this study, a subject must meet all of the following criteria:

6. Diagnosis and history of chronic, moderate-to-severe AD (by the Eichenfield revised criteria of Hanifin and Rajka for at least 3 years before baseline visit.

7. Documented recent history (last 6 months) of eligibility for (local or systemic) treatment with immunosuppressants, biologics or JAK-inhibitors.

8. When applicable, documented recent history (last 6 months) of inadequate response to treatment with topical therapy, immunosuppressants, biologics or JAK-inhibitors.

9. Current treatment can include moisturizers, topical treatment and/or systemic treatments with preferable wash-out (see exclusion criterion #9). On-study treatment is at physician and patient discretion but must include eligibility to starting new systemic treatment.

10. EASI≥7 (moderate-to-severe disease) 11. At least one suitable target lesion at the discretion of the investigator 12. Intention to start treatment with cyclosporine A, dupilumab, tralokinumab, lebrikizumab or a JAK1-inhibitor (abrocitinib or upadacitinib)

For patients with CLE:

Participants must have a diagnosis of CLE, including SCLE, CDLE or LET that fulfil the following:

6. Confirmed CLE diagnosis by clinicopathological correlation. 7. An overall CLE Disease Area and Severity Index Activity (CLASI-A) Score ≥3 without counting any diffuse alopecia or oral ulcers.

8. Intention to start treatment with TCS, hydroxychloroquine or methotrexate (combination or mono-treatment).

If participating in the exploratory study with the skin biopsy: location of the lesion(s) selected for biopsy preferably outside the facial area (possible are e.g., neck, chest, back, limbs, scalp, ear etc.).

For patients with CSU:

6. Diagnosis of CSU (moderate to severe according to international guidelines (Zuberbier et al, 2022)) for ≥3 months and symptomatic disease despite treatment with second generation H1 antihistamines (up to fourfold the approved dose).

7.Patients currently on an antihistamine (up to fourfold the approved dose) must be on a stable dose for at least 2 weeks prior to day 1 and must maintain the same stable dose throughout the treatment period.

8. Intention to start (add-on to antihistamine) treatment of omalizumab, cyclosporine A or BTK inhibitor*. (*when approved and reimbursed in NL)

For patients with HS:

6. Patient with a history of signs and symptoms consistent with moderate-to-severe HS, based on IHS4 score (Zouboulis et al., 2017), for at least 1 year prior to baseline 7. Current treatment can include topical treatment. On-study treatment is at physician and patient discretion but must include eligibility to starting systemic treatment 8. Intention to start treatment with anti-TNF or anti-IL17 (secukinumab, bimekizumab*) *when approved and reimbursed in NL.

For patients with MF:

6. A confirmed diagnosis of CTCL MF type and stage classification via histology or clinicopathological correlation 7. For the stage IA-IIA CTCL patients: at least one patch and/or one plaque lesion is present 8. Intention to start treatment with topical chlormethine, topical corticosteroids or phototherapy (PUVA / UV-B).

For patients with PSO:

6. Diagnosed with chronic plaque psoriasis at least 6 months prior to study participation 7. PASI≥5 with at least one suitable target lesion at the discretion of the investigator 8. Current treatment can include moisturizers, topical treatment and/or systemic treatments with preferable wash-out. On-study treatment is at physician and patient discretion but must include eligibility to starting new systemic treatment 9. Intention to start treatment with biologics: anti-TNF, anti-IL23, anti-IL17 or anti-TYK2

Healthy volunteers:

All healthy volunteers must meet all of the following inclusion criteria:

1. Signed informed consent before any study-mandated procedure.
2. Male or non-pregnant female volunteers, ≥18 years of age
3. Subject is in stable good health as per judgement of the investigator based upon the results of medical history and assessments performed at baseline.
4. No clinically significant skin disease as judged by the investigator.
5. No history of hypertrophic scarring or keloid.
6. Subject is willing to refrain from extensively washing (including bathing, swimming) the skin 12 hours before every study visit.
7. Subject is willing and able to wash out and withhold any topical treatment (prescription and over-the-counter products) in the investigational area for 2 weeks prior to Day 1.
8. Subject is willing to refrain from application of any topical product (e.g. ointments, cream, or washing lotions) on the skin 24 hours prior to every study visit day.
9. Subject is willing and able to wash out any antibiotic therapy for 14 days prior to Day 1.
10. Subject is willing and able to comply with the study protocol.
11. Female participants are willing to not get pregnant from study entry to the last study visit

Exclusion Criteria:

Patients:

1. Have any other relevant skin infection/disease in the treatment area other than the investigated skin disease.
2. Subjects who have received treatment with any non-marketed drug substance (that is, an agent which has not yet been made available for clinical use following registration) within 4 weeks prior to the baseline visit.
3. Any other condition, disease, or known factor that could interfere with the study conduct or the study objectives as per judgement of the investigator. 4. Having received treatments for the investigated skin disease within the following intervals prior to the start of the study is not a strict exclusion criterion since this is a real-world study. However, preferred intervals for washout are as follows:

   * 1 week for topical treatment, e.g. corticosteroids, retinoids, vitamin D analogs, calcineurin inhibitors
   * 4 weeks for phototherapy, e.g. UVB, PUVA, PDT
   * 4 weeks for non-biologic systemic treatment, e.g. retinoids, methotrexate, cyclosporine, JAK inhibitors
   * 8 weeks for radiotherapy or surgery in the treatment area
   * 8 weeks for biologics
   * 3 months for any systemic chemotherapeutical treatment

Disease specific exclusion criteria for patients with CLE:

5. Diagnosed with SLE

Disease specific exclusion criteria for patients with CSU:

5. Treatment with omalizumab within 8 weeks prior to Day 1 6. Urticarial or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary, acquired angioedema or drug-induced (e.g., due to C1 esterase inhibitor deficiency, ACE-inhibitor induced).

Disease specific exclusion criteria for patients with MF:

5. Ongoing uncontrolled active skin infection, other than secondary impetiginized CTCL lesions as judged by the investigator

Disease specific exclusion criteria for patients with PSO:

5. Having primarily erythrodermic, pustular or guttate psoriasis; 6. Having drug-induced psoriasis;

Healthy volunteers:

All healthy volunteers must meet none of the following exclusion criteria:

1. History of immunological abnormality (e.g. immune suppression, severe allergy, or anaphylaxis) that may interfere with study objectives as per judgement of the investigator.
2. History or symptoms of any uncontrolled, significant disease including (but not limited to), a neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder that may interfere with the study objectives as per judgement of the investigator.
3. The use of systemic antibiotic therapy for >2 months in the past 12 months.
4. The use of any immunosuppressive or immunomodulatory therapy within the past 30 days prior to Day 1.

6. Loss or donation of blood over 500mL within three months prior to baseline. Participation in an investigational drug study within 3 months prior to baseline visit or more than 4 times a year.

7. History of alcohol consumption exceeding 5 standard drinks per day on average within 3 months prior to baseline. Alcohol consumption will be prohibited for at least 24 hours preceding each study visit.

8. Positive urine test for drugs or history of abuse at baseline. 9. Exposure to high doses of UV radiation is not permitted within 3 weeks of the first study visit until the end of the study 10. Extreme physical activities are not permitted within 48 hours before each study visit 11. Any other condition, disease, or known factor that could interfere with the study conduct or the study objectives as per judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with six different inflammatory skin diseases (AD, PSO, CLE, HS, CSU, and MF) will be enrolled. Each indication will include multiple treatment groups, with up to 40 patients per group. In total, approximately 120 patients per disease will be studied, except for PSO (4 treatment groups, N=160) and HS (2 treatment groups, N=80), covering a range of disease severities. Patients will be recruited from the local hospital where they receive standard care and will also attend study visits at this location.
  Healthy volunteers will be recruited through the Centre for Human Drug Research.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Lipidomics of the stratum corneum and OLINK | Baseline - month 12
  Tape stripping will be performed on (non-)lesional skin and healthy skin for extraction of lipids for analysis and analysis will be performed using OLINK.
Cutaneous microbiome | Baseline - month 12
  The microbiome is collected by swabbing. The abundance of bacteria is thereafter determined using next-generation sequencing.
Serum biomarkers | Baseline - month 12
  Blood serum will be collected and processed for subsequent biomarker extraction and analysis. The specific biomarkers to be assessed will be determined at a later stage, based on the results of preliminary pilot studies.
Plasma biomarkers | Baseline - month 12
  Blood plasma will be collected and processed for the extraction and analysis of biomarkers. The specific biomarkers to be assessed will be determined at a later stage, based on the results of preliminary pilot studies.
Eczema Area and Severity Index (EASI) | Baseline - month 12
  The Eczema Area and Severity Index (EASI) is a validated clinician-reported outcome measure used to assess the severity and extent of atopic dermatitis. The total EASI score ranges from 0 to 72, with higher scores indicating more severe disease. A score of 0 reflects no disease activity, whereas a score of 72 represents the most severe possible presentation.
  The EASI score will be assessed exclusively in patients diagnosed with atopic dermatitis.
objective Severity Scoring of Atopic Dermatitis (oSCORAD) | Baseline - month 12
  The objective SCORAD (oSCORAD) is a validated clinician-reported outcome measure used to evaluate the severity of atopic dermatitis, focusing on objective clinical signs. The total oSCORAD score ranges from 0 to 83, with higher scores indicating more severe disease. A score of 0 reflects the absence of clinical symptoms, while a score of 83 represents the most severe disease presentation.
  The oSCORAD score will be assessed exclusively in patients diagnosed with atopic dermatitis.
Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) | Baseline - month 12
  The Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) is a clinician-reported outcome measure used to assess the overall severity of atopic dermatitis based on clinical signs. The vIGA-AD score ranges from 0 to 4, with higher scores indicating more severe disease. A score of 0 corresponds to "clear" skin, while a score of 4 represents "severe" disease.
  The vIGA-AD score will be assessed exclusively in patients diagnosed with atopic dermatitis.
Cutaneous LE Disease Area and Severity Index Activity (CLASI-A) | Baseline - month 12
  The Cutaneous Lupus Erythematosus Disease Area and Severity Index - Activity Score (CLASI-A) is a validated clinician-reported outcome measure used to assess the degree of inflammatory disease activity in patients with cutaneous lupus erythematosus. The CLASI-A score ranges from 0 to 70, with higher scores indicating more active and severe skin involvement. A score of 0 reflects no disease activity, while a score of 70 indicates the most severe activity.
  The CLASI-A score will be assessed exclusively in patients diagnosed with cutaneous lupus erythematosus.
Total Sum Score | Baseline - month 12
  The Total Sum Score is a clinician-reported composite outcome measure used to quantify overall disease activity in patients with cutaneous lupus erythematosus and psoriasis. It is calculated by summing the individual scores of predefined clinical signs across affected body regions. The score range depends on the number and weighting of assessed parameters, with higher scores indicating more severe disease activity. A score of 0 reflects no observable disease, whereas the maximum score represents the most severe manifestation based on the scoring algorithm.
  The Total Sum Score will be assessed only in patients diagnosed with cutaneous lupus erythematosus and plaque psoriasis.
The Cutaneous Lupus Activity-Investigator Global Assessment (CLA-IGA) | Baseline - month 12
  The Cutaneous Lupus Activity-Investigator Global Assessment (CLA-IGA) is a validated clinician-reported outcome measure used to assess overall disease activity in patients with cutaneous lupus erythematosus. The scale ranges from 0 to 5, where 0 indicates no disease activity and 5 reflects very severe disease. Higher scores correspond to greater clinical severity.
  The CLA-IGA will be assessed only in patients with cutaneous lupus erythematosus.
International Hidradenitis Suppurativa Severity Score System (IHS4) | Baseline - month 12
  The International Hidradenitis Suppurativa Severity Score System (IHS4) is a validated clinician-reported outcome measure used to assess the severity of hidradenitis suppurativa. The total IHS4 score is calculated based on the number of nodules, abscesses, and draining tunnels, with no fixed maximum but typically ranging from 0 upwards. Higher scores indicate more severe disease activity, while a score of 0 reflects no active disease.
  The IHS4 score will be assessed only in patients with hidradenitis suppurativa.
Modified Severity-Weighted Assessment Tool (mSWAT) | Baseline - month 12
  The Modified Severity-Weighted Assessment Tool (mSWAT) is a clinician-reported outcome measure used to assess the severity and extent of Cutaneous T-Cell Lymphoma, specifically Mycosis Fungoides. The total mSWAT score ranges from 0 to 360, with higher scores indicating more severe disease involvement. A score of 0 reflects no active disease.
  The mSWAT score will be assessed only in patients with Cutaneous T-Cell Lymphoma subtype Mycosis Fungoides.
Cutaneous Lymphoma Activity and Severity Index (CAILS) | Baseline - month 12
  The Cutaneous Lymphoma Activity and Severity Index (CAILS) is a clinician-reported outcome measure used to evaluate disease activity and severity in patients with Cutaneous T-Cell Lymphoma, including Mycosis Fungoides. The total CAILS score ranges from 0 to 70, with higher scores indicating greater disease severity. A score of 0 corresponds to no active disease.
  The CAILS score will be assessed only in patients with Cutaneous T-Cell Lymphoma subtype Mycosis Fungoides.
Psoriasis Area and Severity Index (PASI) | Baseline - month 12
  The Psoriasis Area and Severity Index (PASI) is a validated clinician-reported outcome measure used to assess the severity and extent of plaque psoriasis. The total PASI score ranges from 0 to 72, with higher scores indicating more severe disease. A score of 0 represents no psoriasis involvement.
  The PASI score will be assessed only in patients with psoriasis.
Physician Global Assessment (PGA) | Baseline - month 12
  The Physician Global Assessment (PGA) for Psoriasis is a validated clinician-reported outcome measure used to assess the overall severity of psoriasis, including all clinical forms. The PGA score typically ranges from 0 to 6, depending on the specific scale used, with higher scores indicating more severe disease. A score of 0 represents clear skin with no signs of psoriasis.
  The PGA score will be assessed only in patients with psoriasis.
Body Surface Area (BSA) | Baseline - month 12
  The Body Surface Area (BSA) is a clinician-reported measure used to estimate the percentage of the body affected by psoriasis. The score ranges from 0% to 100%, where 0% indicates no skin involvement and 100% represents the entire body surface affected. Higher BSA values correspond to more extensive disease.
  The BSA will be assessed only in patients with psoriasis.
Psoriasis Area and Severity Index - High Discrimination (PASI-HD) | Baseline - month 12
  The Psoriasis Area and Severity Index - High Discrimination (PASI-HD) is a clinician-reported outcome measure designed to provide enhanced sensitivity and precision in assessing the severity and extent of psoriasis. The score ranges from 0 to 72, where 0 indicates no disease activity and 72 represents the most severe possible presentation. Higher scores correspond to more severe disease.
  The PASI-HD will be assessed only in patients with psoriasis.

SECONDARY OUTCOMES:
User experience and subjective burden questionnaire | Baseline, month 6
  Measures the user experience and subjective burden of the different assessments performed in this study.
Patient reported outcomes | Baseline - month 12
  Patients will be asked to report on the impact of their skin disease on different aspects of their lives, with the following questionnaires: DLQI, TSQM, HADS< NRS pruritus and burning sensation/pain, 5-D itch scale, ISDL, ISBQ, PSWQ, ISDL, expectancies and avoidance behaviour, G-EEE, SQSQ-S, DS-14. The following questionnaires are optional: PSS, P-scale short, and SEMCD. The following disease specific patient reported outcomes are measured: RECAP, POEM, AAS7, UAS7, UCT, HiSQoL.
Skin barrier function by Electrical Impedance Spectroscopy (EIS) | Baseline - month 12
  The barrier status by trans epidermal water loss of (non-)lesional skin and healthy skin will be determined using EIS.
Line-Field Confocal Optical Coherence Tomography (LC-OCT) | Baseline - month 12
  LC-OCT is a non-invasive optical imaging technique based on a combination of the optical principles of optical coherence tomography and reflectance confocal microscopy with line-field illumination, which can generate cell-resolved images of the skin, in vivo, in vertical section, horizontal section and in three dimensions.
Laser Speckle Contrast Imaging (LSCI) | Baseline - month 12
  The cutaneous microcirculation of (non-)lesional skin sites and healthy skin will be monitored over a 40 second timespan with a laser speckle contrast imager.
3D Multispectral imaging | Baseline - month 12
  The redness and superficial morphology of (non-)lesional skin sites and healthy skin will be determined using a 3D multispectral imaging system.
Colorimetry | Baseline - month 12
  The redness and surface characteristics of (non-)lesional and healthy skin will be assessed using a colorimetry device that quantitatively measures skin color parameters, including erythema, based on reflected light.
Skin punch biopsies | Baseline, month 3
  Skin punch biopsies (4mm) will be taken from (non-)lesional skin and healthy for histology, tissue mass cytometry (CyTOF) and RNA-sequencing analysis.
Patient genotyping | Baseline
  A whole blood sample will be used to scan for common mutations in genes implicated in psoriasis using next-generation sequencing.
Activity Tracking Sleep | Baseline - month 6
  Subjects are requested to wear a smartwatch at all times which register sleep (hrs, minutes, seconds of rest)
Activity Tracking Steps | Baseline - month 6
  Subjects are requested to wear a smartwatch at all times which register steps (amount of steps taken)
Activity Tracking Heartrate | Baseline - month 6
  Subjects are requested to wear a smartwatch at all times which heart rate (beats per minute)
Blood sampling for RNAsequencing | Baseline, month 3
  Blood will be drawn during using a venipuncture during visits and analyzed with RNAsequencing.
Dermatology Life Quality Index (DLQI) | Baseline - month 12
  The Dermatology Life Quality Index (DLQI) is a validated patient-reported outcome measure that assesses the impact of skin diseases on patients' quality of life over the previous week. The total DLQI score ranges from 0 to 30, with higher scores indicating greater impairment in quality of life. A score of 0 reflects no impact, whereas 30 represents the most severe impact on quality of life.
  The DLQI will be assessed in all patients across the included skin disease cohorts.
Treatment Satisfaction Questionnaire for Medication (TSQM) | Month 3 - month 12
  The Treatment Satisfaction Questionnaire for Medication (TSQM) is a validated patient-reported outcome measure designed to assess patients' satisfaction with their medication. The TSQM evaluates multiple domains including effectiveness, side effects, convenience, and overall satisfaction. Scores for each domain range from 0 to 100, with higher scores indicating greater satisfaction.
  The TSQM will be assessed in all patients across the included skin disease cohorts.
Hospital Anxiety and Depression Scale (HADS) | Baseline - month 12
  The Hospital Anxiety and Depression Scale (HADS) is a validated patient-reported outcome measure used to assess levels of anxiety and depression symptoms. It consists of two subscales: Anxiety (HADS-A) and Depression (HADS-D), each ranging from 0 to 21. Higher scores indicate greater severity of anxiety or depression symptoms.
  The HADS will be assessed in all patients across the included skin disease cohorts.
Numerical Rating Scale (NRS) for Pruritus and Burning Sensation/Pain | Baseline - month 12
  The Numerical Rating Scale (NRS) for Pruritus and Burning Sensation/Pain are validated patient-reported outcome measures used to assess the intensity of itch and burning pain, respectively. Both scales range from 0 to 10, where 0 indicates no symptom and 10 represents the worst imaginable symptom. Higher scores correspond to greater symptom severity.
  The NRS for pruritus and burning sensation/pain will be assessed in all patients across the included skin disease cohorts.
5-D Itch Scale | Baseline - month 12
  The 5-D Itch Scale is a patient-reported outcome measure designed to assess the multidimensional impact of pruritus (itching). It evaluates five domains: Duration, Degree, Direction, Disability, and Distribution of itch. The total score ranges from 5 to 25, with higher scores indicating greater severity and impact of itch. A score of 5 reflects no itch symptoms, whereas 25 represents the most severe and disabling itch experience.
  The 5-D Itch Scale will be assessed in all patients.
Chronic Skin Disease on Daily Life (ISDL) | Baseline - month 12
  The Chronic Skin Disease on Daily Life (ISDL) is a patient-reported outcome measure designed to evaluate the impact of chronic skin diseases on patients' daily lives. The total score ranges from 0 to 40, with higher scores indicating a greater negative impact on daily functioning and quality of life. A score of 0 reflects no impact, while 40 represents the most severe impairment.
  The ISDL will be assessed in all patients.
Itch Severity and Burden Questionnaire (ISBQ) | Baseline - month 12
  The Itch Severity and Burden Questionnaire (ISBQ) is a validated patient-reported outcome measure designed to assess the psychosocial burden and emotional impact of chronic itch. The total score ranges from 0 to 20, with higher scores reflecting a greater negative impact on emotional wellbeing and daily functioning. A score of 0 indicates no emotional burden, while a score of 20 indicates a very high burden related to chronic itch.
  The ISBQ will be assessed in all patients.
Penn State Worry Questionnaire (PSWQ) | Baseline - month 12
  The Penn State Worry Questionnaire (PSWQ) is a validated patient-reported outcome measure designed to assess the tendency toward excessive, uncontrollable, and generalized worry, which is a key feature of generalized anxiety disorder but may also occur in other chronic conditions.
  The total PSWQ score ranges from 16 to 80, with higher scores indicating greater levels of pathological worry. A score of 16 reflects minimal worry, while a score of 80 reflects a high tendency to worry excessively.
  The PSWQ will be assessed in all patients.
Impact of Chronic Skin Disease on Daily Life (ISDL) | Baseline - month 12
  The Impact of Chronic Skin Disease on Daily Life (ISDL) is a validated patient-reported outcome measure specifically designed to assess the impact of chronic skin conditions on various aspects of daily functioning and quality of life.
  The ISDL consists of multiple domains, including symptoms, emotional burden, daily activities, social functioning, and treatment-related burden. The total score ranges from 0 to 100, with higher scores indicating a greater impact and thus a worse outcome.
  The ISDL will be assessed in all patients.
Expectancies and and avoidance behaviour (G-EEE) | Baseline - month 12
  The Expectancies and Avoidance Behaviour Questionnaire (G-EEE) is a validated patient-reported outcome measure used to assess symptom-related expectancies and avoidance behaviour in individuals with chronic skin conditions. The total score reflects the degree to which patients expect their symptoms to worsen due to certain triggers (e.g. scratching, sweating, stress) and the extent to which they engage in avoidance behaviour as a result. Higher scores indicate stronger avoidance behaviour and more negative symptom-related expectancies. The G-EEE will be assessed in all patient groups.
Social Sensory Processing Questionnaire - Short Form (SPSQ-S) | Baseline - month 12
  The Social Sensory Processing Questionnaire - Short Form (SPSQ-S) is a patient-reported outcome measure designed to assess individual sensitivity to sensory stimuli in social environments. It evaluates how patients perceive and react to social sensory input that may cause discomfort or stress. The questionnaire consists of a series of items scored on a Likert scale, with higher scores indicating greater sensitivity. The SPSQ-S will be assessed in all patient groups.
Type D Personality Scale (DS-14) | Baseline - month 12
  The Type D Personality Scale (DS-14) is a self-reported questionnaire used to identify the presence of a distressed personality type, characterized by high levels of negative affectivity and social inhibition. It consists of 14 items scored on a Likert scale, with higher scores indicating stronger Type D personality traits. The DS-14 will be assessed in all patient groups.
Perceived Stress Scale (PSS) | Baseline - month 12
  The Perceived Stress Scale (PSS) is a self-reported questionnaire designed to measure the perception of stress. It assesses how unpredictable, uncontrollable, and overloaded respondents find their lives. The PSS consists of 10 items scored on a Likert scale, with higher scores indicating higher perceived stress levels. The PSS will be assessed in all patient groups.
P-Scale Short | Baseline - month 12
  The P-Scale Short is a self-reported questionnaire measuring perceived stigma related to chronic illness. It consists of a brief set of items, with higher scores indicating greater experienced stigma. The P-Scale Short will be assessed in all patient groups.
Self-Efficacy for Managing Chronic Disease (SEMCD) scale | Baseline - month 12
  The Self-Efficacy for Managing Chronic Disease (SEMCD) scale is a validated patient-reported outcome measure designed to assess an individual's confidence in their ability to manage symptoms, maintain function, and cope with the emotional and social consequences of chronic diseases. The SEMCD typically consists of multiple items rated on a numerical scale, with higher scores indicating greater self-efficacy and perceived ability to control one's chronic condition. This measure is important for understanding patient empowerment and adherence to treatment plans. The SEMCD will be assessed in all patient groups included in the study.
Recap of Atopic Eczema (RECAP) | Baseline - month 12
  The Recap of Atopic Eczema (RECAP) is a validated patient-reported outcome measure designed to assess disease control over the past week in patients with atopic dermatitis. It consists of a concise set of questions that capture symptoms, impact on daily life, and treatment effectiveness. Scores range from 0 to 30, with higher scores indicating poorer disease control. The RECAP will be assessed only in patients with atopic dermatitis.
Patient-Oriented Eczema Measure (POEM) | Baseline - month 12
  The Patient-Oriented Eczema Measure (POEM) is a validated patient-reported outcome measure used to assess the severity of atopic dermatitis symptoms over the past week. The questionnaire consists of seven items addressing the frequency of key symptoms such as itching, sleep disturbance, and skin dryness. POEM scores range from 0 to 28, with higher scores indicating more severe disease symptoms. The POEM will be assessed only in patients with atopic dermatitis.
Angioedema Activity Score over 7 days (AAS7) | Baseline - month 12
  The Angioedema Activity Score over 7 days (AAS7) is a validated patient-reported outcome measure that captures the severity and frequency of angioedema symptoms during the preceding week. Scores range from 0 to 105, with higher scores indicating greater disease activity and symptom burden. The AAS7 is used exclusively in patients with chronic spontaneous urticaria (CSU) who experience angioedema to monitor short-term disease activity and treatment response.
Urticaria Activity Score over 7 days (UAS7) | Baseline - month 12
  The Urticaria Activity Score over 7 days (UAS7) is a validated patient-reported outcome measure used to assess the severity and frequency of urticaria symptoms-specifically wheals (hives) and pruritus (itch)-over the previous week. Scores range from 0 to 42, with higher scores reflecting more severe disease activity. The UAS7 is applied exclusively in patients with chronic spontaneous urticaria (CSU) to monitor disease burden and evaluate treatment response.
Urticaria Control Test (UCT) | Baseline - month 12
  The Urticaria Control Test (UCT) is a validated patient-reported outcome measure used to assess disease control in patients with chronic spontaneous urticaria (CSU). The total UCT score ranges from 0 to 16, with higher scores indicating better disease control. This questionnaire is used exclusively in patients with CSU to monitor treatment response and disease management over time.
Hidradenitis Suppurativa Quality of Life (HiSQoL) | Baseline - month 12
  The Hidradenitis Suppurativa Quality of Life (HiSQoL) questionnaire is a validated patient-reported outcome measure designed to assess the impact of hidradenitis suppurativa (HS) on patients' quality of life. The total HiSQoL score ranges from 0 to 66, with higher scores indicating greater impairment and worse quality of life. The questionnaire is specifically used in patients with HS to evaluate the burden of disease and monitor changes over time.

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Leiden University Medical Center, Leiden, South Holland
  - Centre for Human Drug Research, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided